CLINICAL TRIAL: NCT01379534
Title: A Phase II, Open-label, Single-arm, Non-randomized, Multi-center Study to Evaluate the Efficacy of Oral TKI258 as Second-line Therapy in Patients With Either FGFR2 Mutated or Wild-type Advanced and/or Metastatic Endometrial Cancer
Brief Title: A Phase II Study to Evaluate the Efficacy of TKI258 for the Treatment of Patients With FGFR2 Mutated or Wild-type Advanced and/or Metastatic Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2211; 2011-000266-35 (EudraCT Number)
Record Dates: First submitted 2011-06-06; First posted 2011-06-23 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Solid Tumors and Advanced Endometrial Cancer; Endometrial Cancer; Second-line Treatment; VEGF
Keywords: Solid tumors,; advanced endometrial cancer,; Endometrial Cancer,; Second-line treatment,; VEGF,; Neoplasms,; Endometrial Neoplasms,; Uterine Neoplasms,; Female Genital Neoplasms,; Cancer,; Carcinoma,; Uterine Diseases,; Female Genital Diseases,; Tumors,; Oral Administration,; Capsules,; Tablets,; CHIR258,; CHIR-258,; CHIR 258,; TKI258,; TKI-258,; TKI 258
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms; Uterine Neoplasms; Genital Neoplasms, Female; Carcinoma; Uterine Diseases; Genital Diseases, Female | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

ARMS (1):
- TKI258 (Experimental): 1 treatment arm (single agent TKI258), with patients classified into 2 groups based on their FGFR2 mutation status
  Interventions: Drug: TKI258

INTERVENTIONS:
Drug: TKI258
  Other Names: dovitinib

SUMMARY:
This is a prospective, multi-center, open-label, single-arm, non-randomized, Phase II study to evaluate the efficacy and safety of TKI258 as second-line therapy in patients with either FGFR2 mutated or wild-type advanced and/or metastatic endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of advanced and/or metastatic endometrial cancer with available tissue specimen (either archival tissue or fixed fresh biopsy)
* Female patients ≥ 18 years old
* Documented radiologically confirmed progression of disease after prior first-line treatment evidence of progressive disease
* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2
* At least one measurable lesion as per RECIST

Exclusion Criteria:

* Previous treatment with an FGFR inhibitor
* More than one line of treatment for advanced or metastatic disease
* Patients with uterine sarcomas, adenosarcoma, and malignant Mullerian tumors
* Patients with isolated recurrences (vaginal, pelvic, or para-aortic) potentially curative with radiation therapy or surgery
* Known central nervous system (CNS) metastases
* Malignancy within 3 years of study enrollment Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (44):
- United States (21):
  - University of South Alabama / Mitchell Cancer Institute Univ South Alabama, Mobile, Alabama
  - St. Jude Heritage Medical Group St Jude, Fullerton, California
  - USC/Kenneth Norris Comprehensive Cancer Center USC 2, Los Angeles, California
  - Cedars Sinai Medical Center TKI258A2211 (SC), Los Angeles, California
  - University of California at Los Angeles UCLA 3, Los Angeles, California
  - Rocky Mountain Cancer Centers Dept. of Rocky Mountain Cancer, Greenwood Village, Colorado
  - Florida Hospital Cancer Institute FL Hosp, Orlando, Florida
  - Indiana University Health Goshen Center for Cancer IU Simon Cancer, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics SC, Iowa City, Iowa
  - Dana Farber Cancer Institute SC, Boston, Massachusetts
  - Southeast Nebraska Oncology Cancer Center, Lincoln, Nebraska
  - Hope A Woman's Cancer Center, Asheville, North Carolina
  - Duke University Medical Center Duke3, Durham, North Carolina
  - Community Oncology Research Network, Chattanooga, Tennessee
  - The West Clinic SC, Memphis, Tennessee
  - Texas Oncology, P.A. Austin, Bedford, Texas
  - Texas Oncology, P.A. Tex Onc (3), Bedford, Texas
  - Texas Oncology, P.A. SC, Fort Worth, Texas
  - South Texas Oncology and Hematology, PA South Tex Onc, San Antonio, Texas
  - Virginia Oncology Associates VOA - Lake Wright, *see Various Departments*, Virginia
  - Cancer Care Northwest SC, Spokane, Washington
- Brazil (3):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
- Italy (6):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Candiolo, TO
- Novartis Investigative Site, Grafton, Auckland, New Zealand
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (7):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Murcia, Murcia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
- United Kingdom (4):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham

REFERENCES:
- [Derived] Konecny GE, Finkler N, Garcia AA, Lorusso D, Lee PS, Rocconi RP, Fong PC, Squires M, Mishra K, Upalawanna A, Wang Y, Kristeleit R. Second-line dovitinib (TKI258) in patients with FGFR2-mutated or FGFR2-non-mutated advanced or metastatic endometrial cancer: a non-randomised, open-label, two-group, two-stage, phase 2 study. Lancet Oncol. 2015 Jun;16(6):686-94. doi: 10.1016/S1470-2045(15)70159-2. Epub 2015 May 13. PMID 25981814

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were treated with TKI258 until disease progression, unacceptable toxicity, death or discontinuation due to any other reason. All participants were followed for at least 30 days after their last dose of study drug for safety assessment.
Pre-assignment Details: If a participant didn't discontinue study drug due to disease progression, death, lost to follow-up or withdrawn consent to post treatment tumor assessment, then tumor assessments continued every 6 weeks until the start of new anti-cancer therapy, disease progression, death, lost to follow-up or withdrawn consent to tumor status follow-up.
Groups:
- FGFR2 (MUT); FGFR2 (WT): Participants were classified into two groups based on mutational status of FGFR2 and all participants were treated with 500 mg of TKI258on a 5 day on / 2 days off dosing regimen for 13 weeks.
Period: Treatment Phase
Arm/Group | FGFR2 (MUT) | FGFR2 (WT)
Started | 22 | 31
Completed | 0 | 0
Not Completed | 22 | 31
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Progressive disease | 13 | 22
Not completed — Adverse Event | 7 | 7
Period: Tumor Assessment Follow-up (f/u) Phase
Arm/Group | FGFR2 (MUT) | FGFR2 (WT)
Started | 4 (All participants discontinued the Treatment Phase. Of these, only 6 qualified for f/u tumor assess..) | 2
Completed | 0 | 0
Not Completed | 4 | 2
Not completed — Death | 0 | 1
Not completed — Progressive disease | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FGFR2 (MUT) | FGFR2 (WT) | Total
Number analyzed (Participants) | 22 | 31 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (10.54) | 64.4 (8.63) | 63.4 (9.45)
Sex/Gender, Customized [Number; unit: Participants] — Females only
  Participants | 22 | 31 | 53

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Rate
Description: The 18-week PFS was defined as the percentage of participants who did not have a progression event at week 18. Participants who progressed, died, had response assessment of unknown (UNK) or discontinued before 18 weeks of observation without progression were counted as "failure". Progressive disease was assessed as per investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Time Frame: up to 18 weeks
Population: Primary endpoint analysis set (PEAS): The PEAS included all participants who received at least one dose of study medication and had measurable disease at baseline as confirmed by a local Investigator.
Measure: Number; unit: Percentage of participants
Arm/Group | FGFR2 (MUT) | FGFR2 (WT)
Number analyzed (Participants) | 22 | 31
Percentage of participants | 31.8 | 29.0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR).
Time Frame: Baseline and every 6 weeks until disease progression, up to 18 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | FGFR2 (MUT) | FGFR2 (WT)
Number analyzed (Participants) | 22 | 31
Percentage of participants | 4.5 | 16.1

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with a best overall response of CR or PR or stable disease (SD).
Time Frame: Baseline and every 6 weeks until disease progression, up to 18 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | FGFR2 (MUT) | FGFR2 (WT)
Number analyzed (Participants) | 22 | 31
Percentage of participants | 63.6 | 51.6

4. Secondary Outcome: Duration of Response (DR)
Description: Duration of response was defined for participants with a CR or PR as the time from the date of the first documented response (CR or PR) to the date of the first documented progression or death due to disease. If a participants did not have a progression event, duration of response was censored at the date of the last adequate tumor assessment before the data analysis cut-off date or the antineoplastic therapy start date or the death date.
Time Frame: up to 18 weeks
Population: This outcome measure was not analyzed. The analysis was not required because there were too few responders.
Arm/Group | FGFR2 (MUT) | FGFR2 (WT)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of treatment to the date of death from any cause. If a participant was not known to have died at the date of analysis cut-off, the OS was censored at the last date of contact.
Time Frame: up to 18 weeks
Population: Full Analysis Set (FAS): The FAS included all participants who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FGFR2 (MUT) | FGFR2 (WT)
Number analyzed (Participants) | 22 | 31
Months | 20.2 [8.2 to 20.2] | 9.3 [6.0 to 15.2]

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause. If a participant did not have an event, PFS was censored at the date of last adequate response assessment before the data analysis cut-off date or the start date of new antineoplastic therapy after study drug discontinuation.
Time Frame: up to 18 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FGFR2 (MUT) | FGFR2 (WT)
Number analyzed (Participants) | 22 | 31
Months | 4.1 [2.6 to 5.5] | 2.7 [1.4 to 6.8]

7. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Deaths
Description: Adverse event monitoring was conducted throughout the study.
Time Frame: up to 30 days after the last dose of study drug, up to 18 weeks
Population: Safety analysis set: The safety set included all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | FGFR2 (MUT) | FGFR2 (WT)
Number analyzed (Participants) | 22 | 31
Participants
  Adverse events (serious and non-serious) | 22 | 31
  Serious adverse events | 10 | 20
  Deaths | 1 | 4

ADVERSE EVENTS:
Arm/Group | FGFR2 (MUT) | FGFR2 (WT)
Serious Adverse Events (participants affected / at risk) | 10/22 | 20/31
Other Adverse Events (participants affected / at risk) | 21/22 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FGFR2 (MUT) (N=22) | FGFR2 (WT) (N=31)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 1
GASTROINTESTINAL ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 3
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 2
PANCREATIC DUCT DILATATION (Gastrointestinal disorders) | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 3
VOMITING (Gastrointestinal disorders) | 2 | 5
FATIGUE (General disorders) | 0 | 1
LOCALISED OEDEMA (General disorders) | 0 | 1
MALAISE (General disorders) | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 2
PYREXIA (General disorders) | 0 | 2
HEPATITIS TOXIC (Hepatobiliary disorders) | 1 | 0
JAUNDICE (Hepatobiliary disorders) | 1 | 0
SEPSIS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 2
UROSEPSIS (Infections and infestations) | 1 | 0
GASTROENTERITIS RADIATION (Injury, poisoning and procedural complications) | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 1
PLATELET COUNT DECREASED (Investigations) | 0 | 1
TRANSAMINASES INCREASED (Investigations) | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 1
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 2
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 | 1
UROGENITAL FISTULA (Renal and urinary disorders) | 0 | 1
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 0 | 2
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 1
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 2
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 | 0
EMBOLISM (Vascular disorders) | 1 | 2
HYPERTENSION (Vascular disorders) | 0 | 2
HYPOTENSION (Vascular disorders) | 0 | 2
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 1
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FGFR2 (MUT) (N=22) | FGFR2 (WT) (N=31)
ANAEMIA (Blood and lymphatic system disorders) | 3 | 10
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 2
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 4
TINNITUS (Ear and labyrinth disorders) | 0 | 2
DRY EYE (Eye disorders) | 2 | 4
EYE DISCHARGE (Eye disorders) | 0 | 2
OCULAR HYPERAEMIA (Eye disorders) | 0 | 3
VISION BLURRED (Eye disorders) | 0 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 6
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 2
CONSTIPATION (Gastrointestinal disorders) | 4 | 6
DIARRHOEA (Gastrointestinal disorders) | 14 | 24
DRY MOUTH (Gastrointestinal disorders) | 3 | 3
DYSPEPSIA (Gastrointestinal disorders) | 4 | 5
FLATULENCE (Gastrointestinal disorders) | 2 | 4
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 2
NAUSEA (Gastrointestinal disorders) | 16 | 21
STOMATITIS (Gastrointestinal disorders) | 1 | 2
VOMITING (Gastrointestinal disorders) | 14 | 21
ASTHENIA (General disorders) | 4 | 5
FATIGUE (General disorders) | 9 | 16
LOCAL SWELLING (General disorders) | 2 | 0
OEDEMA PERIPHERAL (General disorders) | 2 | 4
PAIN (General disorders) | 0 | 6
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2
URINARY TRACT INFECTION (Infections and infestations) | 3 | 3
CONTUSION (Injury, poisoning and procedural complications) | 0 | 2
FALL (Injury, poisoning and procedural complications) | 0 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 | 3
AMYLASE INCREASED (Investigations) | 0 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 2
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 | 8
BLOOD BILIRUBIN INCREASED (Investigations) | 2 | 0
BLOOD CHOLESTEROL INCREASED (Investigations) | 1 | 3
BLOOD CREATININE INCREASED (Investigations) | 3 | 4
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 | 2
LIPASE INCREASED (Investigations) | 2 | 2
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 | 2
PLATELET COUNT DECREASED (Investigations) | 1 | 2
WEIGHT DECREASED (Investigations) | 7 | 5
DECREASED APPETITE (Metabolism and nutrition disorders) | 9 | 9
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 5
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1 | 4
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 5
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 2 | 9
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 | 5
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 4
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 4 | 6
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 5
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 | 2
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 3
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 | 9
DIZZINESS (Nervous system disorders) | 3 | 7
DYSGEUSIA (Nervous system disorders) | 2 | 2
HEADACHE (Nervous system disorders) | 5 | 6
PARAESTHESIA (Nervous system disorders) | 2 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 2
ANXIETY (Psychiatric disorders) | 0 | 2
INSOMNIA (Psychiatric disorders) | 2 | 2
DYSURIA (Renal and urinary disorders) | 0 | 4
PROTEINURIA (Renal and urinary disorders) | 1 | 3
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 1 | 2
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 3 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 6
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 7
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 3
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 2
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 | 2
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 2 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 3
RASH (Skin and subcutaneous tissue disorders) | 9 | 11
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 2
EMBOLISM (Vascular disorders) | 2 | 1
HYPERTENSION (Vascular disorders) | 4 | 8
HYPOTENSION (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.